CLINICAL TRIAL: NCT06143839
Title: VYxeoS Liposomal Italian Observational Study iN the Real Practice
Acronym: VYSION
Status: Completed | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Advice Pharma S.r.l. (Unknown)
Responsible Party: Sponsor
Other Study IDs: JZP351-501
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Myeloid Leukemia With Myelodysplasia-Related Changes; Therapy-Related Acute Myeloid Leukemia
Keywords: JZP351; CPX-351; Vyxeos liposomal; AML; t-related AML; AML-MRC
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Myeloid Leukemia (AML): Participants with newly diagnosed AML-MRC (Acute myeloid leukemia with myelodysplasia-related changes) or t-related AML (Therapy related Acute myeloid leukemia) receiving Vyxeos liposomal as part of their standard of care treatment.
  Interventions: Drug: Vyxeos liposomal

INTERVENTIONS:
Drug: Vyxeos liposomal — Standard of care JZP351 administered intravenously over 90 minutes.
  Other Names: JZP351; CPX-351

SUMMARY:
The study is a prospective, single-arm, non-experimental, observational study in patients in Italy with Acute Myeloid Leukaemia (AML) with myelodysplastic-related changes or therapy related AML initiating treatment with JZP351 (Vyxeos liposomal) in their normal clinical practice.

ELIGIBILITY:
Inclusion criteria:

* Patients newly diagnosed with AML-MRC (Acute myeloid leukemia with myelodysplasia-related changes) or t-related AML (Therapy related Acute myeloid leukemia) following 2016 World Health Organization (WHO) classification.
* Age ≥ 18 years old.
* Patients considered eligible for intensive chemotherapy in the opinion of the treating physician.
* Patients who will initiate the treatment with commercially JZP351 treatment after the Informed Consent Form (ICF) signature. The decision to prescribe JZP351 treatment must have been made prior and regardless of the enrollment of the patient in the study.
* Cardiac ejection fraction ≥ 50% by echocardiography or MUGA (Multi-Gated Acquisition).

Exclusion criteria:

* Prior treatment intended for induction therapy of AML (Acute Myeloid Leukemia).
* Patients with prior cumulative anthracycline exposure of greater than 368 mg/m2 daunorubicin (or equivalent)
* Clinical evidence of active CNS (Central Nervous System) leukemia.
* Patients with active (uncontrolled, metastatic) second malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with t-AML or AML-MRC considered suitable for intensive chemotherapy who will be receiving JZP351 (Vyxeos liposomal) as part of their normal clinical care in Italian hematology centers.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Percentage of participants showing CR/CRi/CRh without MRD at the end of treatment | Up to 24 months
  Percentage of participants showing CR (Complete Remission) / CRi (Complete Response with incomplete platelet or neutrophil recovery) /CRh (Complete Response with partial hematologic recovery) without MRD (measurable residual disease) at the end of treatment. MRD will be assessed via multiparameter flow cytometry.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) after induction phase | Up to 24 months
  ORR is the rate of participants achieving CR, CRi and CRh after induction phase
Percentage of participants showing CR/CRi/CRh without MRD after induction phase | Up to 24 months
  MRD will be assessed via multiparameter flow cytometry.
Percentage of participants showing CR/CRi/CRh without MRD before transplantation | Up to 24 months
  MRD will be assessed via multiparameter flow cytometry.
Overall survival (OS) | Up to 24 months
  Overall survival is date from the start of taking Vyxeos liposomal (JZP351) to the date of reported death due to any cause.
Percentage of participants receiving an Hematopoietic stem-cell transplantation (HSCT) | Up to 24 months
Landmark overall survival (OS) from the time of HSCT | Up to 24 months
Percentage of participants with Adverse Events (AE) | Up to 24 months
  Percentage of participants who experience Grades 1-5 and grade 3-5 adverse events, including AEs of special interest and serious AEs (SAEs), as evaluated by treating physician.
Percentage of participants with a change in fitness status as assessed by Ferrara criteria before HSCT | Up to 24 months
  Ferrara criteria is a list of assessments evaluating whether a participant is eligible for intensive chemotherapy or not.
Percentage of participants with a change in fitness status as assessed by Ferrara criteria at the final treatment visit for patients not eligible for HSCT | Up to 24 months
  Ferrara criteria is a list of assessments evaluating whether a participant is eligible for intensive chemotherapy or not.

CONTACTS AND LOCATIONS:
Locations (24):
- Italy (24):
  - Azienda ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Policlinico Sant'Orsola, Bologna
  - Ospedale di Bolzano, Bolzano
  - Ospedale Busto Arsizio, Busto Arsizio
  - Istituto Oncologico Veneto, Castelfranco Veneto
  - Ospedale Careggi, Florence
  - Policlinico San Martino, Genova
  - Ospedale Vito Fazzi, Lecce
  - Policlinico di Milano Ospedale Maggiore, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Ospedale Cardarelli, Napoli
  - Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Ospedale Civile Santo Spirito, Pescara
  - Ospedale Santa Chiara, Pisa
  - Ospedale di Ravenna, Ravenna
  - Ospedale Bianchi Melacrino Morelli, Reggio Calabria
  - Policlinico Tor Vergata, Roma
  - Ospedale Sant'Eugenio, Roma
  - Policlinico Umberto I, Roma
  - Policlinico Agostino Gemelli, Roma
  - Policlinico Molinette, Torino
  - Ospedale Riuniti Marche Nord, Torrette Ancona
  - Ospedale di Trieste, Trieste

IPD SHARING:
Plan to Share IPD: No